CLINICAL TRIAL: NCT07239687
Title: Comparison of Eleveld and Schnider Models for Target-Controlled Infusion of Propofol in Intensive Care Unit Sedation
Brief Title: A Comparative Study of Eleveld and Schnider Pharmacokinetic Models for Target-Controlled Infusion of Propofol in Sedation of Mechanically Ventilated ICU Patients
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Özdemir Şimşek, Medical resident in anesthesiology, Hacettepe University
Other Study IDs: 2024/15-02 (KA-24022)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Intensive Care Unit Sedation; Sedation; Target Controlled Infusion of Propofol
Keywords: Propofol, Target-Controlled Infusion, Eleveld Model, Schnider Model, ICU, Sedation, BIS, Riker Scale
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Eleveld Model Group: Patients sedated with propofol using the Eleveld pharmacokinetic model via a target-controlled infusion (TCI) system. Sedation will be titrated to maintain a Riker Sedation-Agitation Scale score between 3 and 4 and a Bispectral Index (BIS) value of 60-80. Hemodynamic variables, awakening time, and total propofol dose will be recorded for comparison with the Schnider group.
  Interventions: Drug: propofol; Device: TCI Propofol Injection
- Schnider Model Group: Patients sedated with propofol using the Schnider pharmacokinetic model via a target-controlled infusion (TCI) system. Sedation depth and hemodynamic parameters will be monitored using the same protocol as in the Eleveld group. BIS values, Riker scores, and recovery profiles will be compared to assess pharmacodynamic and clinical performance between models.
  Interventions: Drug: propofol; Device: TCI Propofol Injection

INTERVENTIONS:
Drug: propofol — Propofol will be administered via a target-controlled infusion (TCI) system for sedation of mechanically ventilated ICU patients. Two pharmacokinetic models, Eleveld and Schnider, will be used to guide the infusion. Sedation depth will be titrated to achieve a Riker Sedation-Agitation Scale score between 3 and 4 and a Bispectral Index (BIS) value of 60-80. Hemodynamic parameters, total propofol dose, awakening time, and incidence of delirium will be recorded for comparison between models. No other sedative or hypnotic agents will be used during the study period.
  Other Names: Diprivan
Device: TCI Propofol Injection — Propofol will be administered intravenously via a target-controlled infusion (TCI) system for sedation of mechanically ventilated intensive care unit (ICU) patients. The infusion will be guided by two different pharmacokinetic models - Eleveld and Schnider - assigned to respective patient groups. The TCI device automatically adjusts infusion rates to maintain target effect-site concentrations according to each model. Sedation depth will be titrated to maintain a Riker Sedation-Agitation Scale score of 3-4 and a Bispectral Index (BIS) value between 60 and 80. Hemodynamic variables, awakening time, and delirium incidence will be evaluated to compare clinical performance between the two models.

SUMMARY:
This prospective observational study aims to compare the clinical performance of two target-controlled infusion (TCI) models, Eleveld and Schnider, for propofol sedation in mechanically ventilated intensive care unit (ICU) patients. The study evaluates sedation depth, hemodynamic stability, and recovery profiles using the Bispectral Index (BIS) and Riker Sedation-Agitation Scale. Secondary outcomes include awakening time, total propofol dose, and incidence of delirium after sedation withdrawal. The findings may help identify the most reliable pharmacokinetic model for safe and effective ICU sedation.

ELIGIBILITY:
Inclusion Criteria:

Age over 18 years,

Classified as ASA (American Society of Anesthesiologists physical status) class I-IV,

Being monitored in the Anesthesiology and Reanimation Intensive Care Unit of Hacettepe University Faculty of Medicine Hospital,

Availability of necessary data (medical history, laboratory results, etc.) for analysis,

Hemodynamic stability -

Exclusion Criteria:Patients who refused to participate in the study or did not provide legal consent,

Patients with an ASA (American Society of Anesthesiologists physical status) classification greater than IV,

Transition to an alternative sedation method during the study,

Contraindication to propofol infusion (e.g., propofol anaphylaxis, lipid metabolism disorders),

Patients whose sedation level could not be clinically assessed due to neurological or neurodegenerative diseases,

Patients expected to require sedation for more than 72 hours (to reduce the risk of propofol infusion syndrome)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18 years or older) admitted to the intensive care unit (ICU) who require continuous sedation with propofol during mechanical ventilation. All patients are hemodynamically stable at the time of sedation initiation and are expected to require sedation for at least 24 hours. Patients are managed according to standard ICU protocols, including daily sedation assessments and monitoring with the Bispectral Index (BIS) and Riker Sedation-Agitation Scale.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Sedation Depth Control Measured by BIS Values | During the sedation period (up to 72 hours)
  Comparison of the accuracy and stability of target-controlled infusion (TCI) sedation between the Eleveld and Schnider pharmacokinetic models in mechanically ventilated ICU patients. Sedation depth will be assessed by Bispectral Index (BIS) monitoring and maintained between 60 and 80. The mean absolute deviation of BIS from target range will be calculated to evaluate model performance
Accuracy of Sedation Depth Control Measured by BIS Values | During the sedation period (up to 72 hours)
  Comparison of the accuracy and stability of target-controlled infusion (TCI) sedation between the Eleveld and Schnider pharmacokinetic models in mechanically ventilated ICU patients. Sedation depth will be assessed by Bispectral Index (BIS) monitoring and maintained between 60 and 80. The mean absolute deviation of BIS from target range will be calculated to evaluate model performance.

SECONDARY OUTCOMES:
Proportion of Time Within Target Sedation Range (Riker Score 3-4) | During the sedation period (up to 72 hours)
  Percentage of total sedation time during which patients remained within the target Riker Sedation-Agitation Scale (SAS) range of 3-4, comparing the Eleveld and Schnider TCI propofol models.

CONTACTS AND LOCATIONS:
Overall Officials: BASAK AKCA, Associate Professor, Study Director — Hacettepe University Faculty of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schnider TW, Minto CF, Shafer SL, Gambus PL, Andresen C, Goodale DB, Youngs EJ. The influence of age on propofol pharmacodynamics. Anesthesiology. 1999 Jun;90(6):1502-16. doi: 10.1097/00000542-199906000-00003. PMID 10360845

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT07239687/Prot_SAP_000.pdf